CLINICAL TRIAL: NCT02002169
Title: Hemodialysis Infection Prevention Using Polysporin Ointment With Shower Technique in Satellite Centres (HIPPO SAT) Pilot Study
Brief Title: Hemodialysis Infection Prevention Using Polysporin Ointment With Shower Technique in Satellite Centres Pilot Study
Acronym: HIPPO-SAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Scarborough General Hospital (Other); London Health Sciences Centre (Other); Trillium Health Centre (Other); York Central Hospital, Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REB 12-0404-AE
Record Dates: First submitted 2013-11-28; First posted 2013-12-05 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: End Stage Renal Failure on Dialysis
Keywords: Catheter Related Bacteremia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Shower Technique Protocol (STP) (Experimental): Participants will be given a minimum 30 minute personalized educational session by the study coordinator. They will be taught safe and clean techniques for showering with their CVC. If the participant passes the Shower Technique Test, they will be provided a pamphlet on the STP, not to be shared with other participants, to be kept as a reference and placed in their bathroom/household. They will also be given the necessary supplies for the STP.
  Interventions: Other: Shower Technique Protocol; Other: Standard CVC Care
- Standard CVC care (Active Comparator): Standard CVC Care consists of cleansing with chlorhexidine 2% or povidone (if allergic to chlorhexidine) at the CVC exit site by trained HD nurses followed by placement of a dry gauze dressing by the HD nurse 1x/week or when clinically indicated. In order to participate in the standard CVC care arm, participating sites must have in their policy that it is trained HD nurses who will apply the Polysporin Triple Ointment after standard cleansing with chlorhexidine 2% or povidone during HD, according to guideline recommendations or as per hospital patient care standards and nursing regulations.
  Interventions: Other: Standard CVC Care

INTERVENTIONS:
Other: Shower Technique Protocol — Video and educational pamphlets of the STP will be used to assist in training participants randomized to this intervention. The participant must successfully demonstrate the STP on a training mannequin and be deemed by the study coordinator as ready to independently and correctly perform it before proceeding.
  Arms: Shower Technique Protocol (STP)
Other: Standard CVC Care — Nuanced differences may be present at participating units; however, the key components of the intervention are 1) HD nurse delivery of CVC care 2) chlorhexidine or povidone cleansing 3) dry gauze dressing 4) standardized frequency. For both STP and control arms, participants whose HD centre uses polysporin triple ointment as part of standard CVC care will continue to have it applied as per program policy.

SUMMARY:
Background: The investigators developed a Shower Technique protocol (STP) for hemodialysis (HD) patients with healed central venous catheter (CVC) exit sites, designed to permit showering but not increase infection risk.

Research question: Is it feasible to conduct a randomized control trial comparing the rate of CVC related bacteremia (CRB) in adult satellite HD patients using STP versus standard CVC care alone with 6 month follow up? Study Design: This pilot study is a multi-centre randomized control trial. Eligible participants will be randomized to STP versus standard care after meeting predefined criteria to confirm healed tunneled CVC exit site.

Primary Outcome: Feasibility will be determined based on 5 outcome measures: accuracy of the CRB rate documentation in the satellite setting, percentage of patients screened, recruited, educated successfully in the STP (intervention arm), and aspects of STP (% of contaminated patients in the control arm).

Study Setting: In satellite units affiliated with 2 academic and 3 community centres in south central Ontario, Canada.

Patient Population: Adult satellite HD patients dialyzing via CVC with healed CVC exit sites.

Intervention: STP and standard CVC care; or Control: standard CVC care; Analysis: Each measure of feasibility has its statistical threshold for success. If the threshold is reached in 4 of the 5 measures, the full HIPPO SAT study will be deemed feasible.

Discussion: A pilot feasibility study of the larger study is critical due to the potential challenges associated with recruitment, compliance and contamination.

DETAILED DESCRIPTION:
CVC related infections are associated with increased morbidity and hospitalization rates, high treatment costs, and poor survival compared to use of an arteriovenous access. To prevent infection, patients should preserve the integrity and dryness of their CVC dressings. Showering should be avoided, as it is difficult to attain full protective coverage of the exit site using dressings and barriers. Wet dressings place patients at increased infection risk, especially if their CVC exit site is not fully healed. However, in a survey of 274 CVC dependent HD patients, 64% indicated that the recommended prohibition to shower was moderately to extremely inconvenient and reduced their quality of life. Additionally 77% of patients admitted to showering at least once while they had a CVC.

While submersion of the CVC in water is discouraged by clinical practice guidelines, they also state that if precautions can be taken to reduce the likelihood of bacterial CVC entry then showering may be acceptable. However, this guidance is opinion based with no evidence to support specific precautions. Thus, to address the patients' desire to shower safely, at least 2 separate dialysis facilities in Ontario, Canada have developed a showering procedure as an alternative method of CVC care. Preliminary data from a small proof-of-concept study of 65 patients suggests acceptable CRB rates (0.46/1000 CVC days) using such showering procedures. The study was conducted in satellite HD units on a select population of patients who were infection-free for 6 months using the same CVC. Satellite units offer dialysis in an outpatient setting for those patients who are stable and require less intensive care than in-centre patients. The satellite HD population is typically younger and healthier, and likely more able to perform showering procedures than in-centre patients. With increasing patients in satellite HD, it is crucial that a pragmatic, yet effective, prophylactic CVC infection strategy be formally tested and established for this setting.

Following the proof-of-concept study, nephrologists, vascular access coordinators, and HD centres from five dialysis centres across Ontario, collaborated to create a formal Shower Technique Protocol (STP) which includes chlorhexidine applicators after showering to minimize the risk of bacterial entry at the CVC exit site. STP is designed specifically for patients with a fully endothelialized CVC tunnel and healed exit site. Participants allocated to STP are able to shower and change their dressing up to 3 times per week. Prior to more widespread implementation of the STP, it is critical to determine whether it is safe for use in patients with healed CVC exit sites. In other words, to confirm that CRB rates in patients using STP are not greater than the CRB rates in patients using the gold standard of CVC care. It is unknown whether using the STP improves patient satisfaction with their CVC care.

ELIGIBILITY:
Inclusion Criteria

* Informed written consent obtained (English speaking)
* Age >18 years
* Requires a CVC as the vascular access: a) end stage kidney disease without a functioning surgically created access; b) end stage kidney disease whose peritoneal dialysis problems require transfer to HD for an anticipated prolonged period
* Passed 2/3 tests of CVC exit site healing (see below)
* Must be willing and able to take a shower as the standard form of body cleansing if randomized to STP
* Trisodium citrate (4%) as standard CVC locking solution
* CVC has been in situ for > 6 weeks

Exclusion criteria

* Acute kidney failure, likely to be reversible with recovery of renal function
* Non-Tunneled CVC
* Antibiotic use by any route in the week prior to enrolling in the study, including intranasal mupirocin
* On immunosuppressant therapy
* Use of the CVC for purposes other than access for hemodialysis
* Involvement in another interventional study related to their vascular access
* CVC or patient life expectancy <6 months (e.g. active malignancy; serious comorbidity such as hepatic failure)
* Routine use of tissue plasminogen activator or antibiotic as a locking solution
* CVC insertion in location other than the neck/chest region (IJ or subclavian acceptable)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-07 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Primary Feasibility Measure of the HIPPO SAT trial: Defined by 5 outcomes | 6 months
  Outcome Measures of Feasibility
  1. The level of agreement between the date the nurse contacts the coordinator to inform them of a suspected infection and the date the culture was sent to the lab from the HD unit
  2. The percentage of eligible patients who consent to participate in each participating satellite unit
  3. The percentage of satellite HD patients with CVCs who are screened for eligibility
  4. The percentage of patients in the Shower Technique arm passing the shower technique test at 3 and 6 months
  5. The percentage of patients in the control arm who are contaminated i.e. using aspects of the STP such as chlorhexidine swabs at home at the exit site which they were not using at baseline

SECONDARY OUTCOMES:
Secondary Feasibility Outcome: The change in Vascular Access Questionnaire (VAQ) score over time using the Shower Technique protocol compared to standard care. | 6 months
  The VAQ is a measure of patient satisfaction with their vascular access that is previously un validated in this population
Secondary Feasibility Outcome: The level agreement between the Deep Breath and CVC Seal tests and the blinded photo test | After consent and prior to randomization
  Once written consent is obtained, the participant will undergo formal testing for CVC exit site healing. The tests of CVC exit site healing are as follows: 1) Deep Breath Stability Test measures the migration of the CVC as marked by a 2 cm indicator on the CVC from the skin at CVC exit. There should be < 3 mm movement between complete exhalation and inhalation; 2) CVC Seal Test is a visual inspection against an objective checklist to determine healing; and 3) Blinded Photo Test where two photos are taken of the CVC exit site to be evaluated for healing by independent blinded trained assessors. Both assessors must agree that the exit site is healed to pass the test.

OTHER OUTCOMES:
Primary Clinical Outcome Measure: The number of confirmed catheter related bacteremia per 1,000 access days | 6 months
  Each catheter related bacteremia will be confirmed by the Hemodialysis Infection Control Subcommittee committee at Toronto General Hospital
Secondary Clinical Outcome: Patient satisfaction will be measured by the Vascular Access Questionnaire score | Baseline, 3 and 6 months
Secondary Clinical Objective: The mean cost per patient of using the Shower Technique protocol versus standard care | 6 months
  The frequency and type of dressings, as well as the frequency of dressing changes by nurse and patient will be prospectively recorded for all patients in the study
Tertiary Clinical Objective: Proportions of patients with CRB, CVC related infection and tunnel infection | 6 months
  As defined by the Health Canada, determined by the independent event adjudication committee (Hemodialysis Infection Control Subcommittee using the "Suspected CVC related infection outcome reporting form" completed by the nurse at the time infection is suspected, the lab reports, and a detailed chart review following a suspected infection for any related CVC removal, hospitalization, and death.
Tertiary Clinical Objective: The number of days to this first CVC related infection from the date of randomization | 6 months
Tertiary Clinical Objective: The rate of CVC removal due CVC related infection as recorded in the vascular access record | 6 months
Tertiary Clinical Objective: The number of days in hospital due to CVC related infection | 6 months
Tertiary Clinical Objective: The proportion of patients who die from CVC related infection | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Charmaine Lok, MD, MSc, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada